CLINICAL TRIAL: NCT04494685
Title: Effects of Robotic Rehabilitation in Post-Stroke Patients: A Randomized Controlled Trial
Brief Title: Effects of Robotic Rehabilitation in Post-Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Rodrigo Della Méa Plentz, PhD, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Stroke_ERIGO
Record Dates: First submitted 2020-05-29; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Stroke
Keywords: Stroke; Robotics; Electric stimulation
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic rehabilitation (Experimental): Robotic rehabilitation with Erigo® equipment (Hocoma, Volketswil, Switzerland).
  Interventions: Device: Intervention group (Robotic rehabilitation)
- Conventional physiotherapy (Active Comparator): The protocol will be based on lower limb exercises, aiming at maintaining and gaining muscle strength through passive, assisted or active mobilization, when possible, on the affected side.
  Interventions: Other: Control group (Conventional physiotherapy)

INTERVENTIONS:
Device: Intervention group (Robotic rehabilitation) — Robotic rehabilitation with Erigo® equipment (Hocoma, Volketswil, Switzerland). The training protocol has a progression of the board inclination up to 90º associated with flexion/extension movements of the knees and hips, with time evolution of up to 40 minutes. Such equipment is associated with electrostimulation of the quadriceps, hamstrings, sural triceps and anterior tibialis.
  Other Names: Erigo®
  Arms: Robotic rehabilitation
Other: Control group (Conventional physiotherapy) — Knee and hip flexion and extension movements, hip adduction, and abduction, respecting the articular physiology of each joint. Weight transfer will also be performed in the sitting and standing position, mini squat, and gait training. All exercises will have a total of 10 repetitions in three sets. In the end, stretching of the upper and lower limbs will be performed.
  Arms: Conventional physiotherapy

SUMMARY:
This study aims to evaluate the effect of robotic rehabilitation through training on a robot-assisted orthostatic board and neuromuscular electrical stimulation (NMES) on functionality in post-stroke patients. In this randomized controlled trial the patients will be allocated to a control group (which will receive conventional physiotherapy) or or to intervention group (which will receive conventional physiotherapy and robotic rehabilitation). Interventions will occur every day in the hospital phase and three times/week after discharge, totaling 18 sessions.The groups will be evaluated prior to any physiotherapy intervention, in the 10h session and at the end of six weeks of treatment (or 18 sessions).The following outcomes will be measured: functionality, peripheral muscle strength, muscle architecture and echogenicity, spasticity, cardiorespiratory repercussions, mobility, disability and dependence, quality of life and time of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of ischemic stroke, in the subacute phase (after 48 hours);
* To present hemiparesis or muscle weakness defined by the Medical Research Council (MRC) score;
* To understand simple commands and being able to report signs of discomfort.

Exclusion Criteria:

* Severe psychomotor agitation;
* Recent acute myocardial infarction (24 hours) and/or uncontrolled arrhythmias;
* Intracranial hypertension (PIC> 20mmHg);
* Uncontrolled hypertension (PAS> 230 mmHg and PAD> 120 mmHg) or PAM <60 mmHg;
* Decompensated heart failure;
* To present important hemodynamic changes during training;
* Peripheral vascular disease in the lower limb such as untreated deep vein thrombosis;
* Unconsolidated fractures or severe joint pain;
* Feverish state;
* Smokers;
* Epidermal lesions on the thighs that make it impossible to place self-adhesive electrodes for electrical stimulation;
* Pre-existing neuromuscular disease;
* Signs of rhabdomyolysis;
* Pregnancy.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Functionality | Baseline, after 3 weeks and after 6 weeks
  The change in functionality will be assessed using the Fugl-Meyer Scale. This scale consists of six domains: range of motion, pain, sensitivity, motor function of the upper and lower extremities, balance, coordination and speed. The score for each item ranges from 0 to 2, where 0 = cannot be performed; 1 = partially accomplished; 2 = completely accomplished. The total score ranges from 0 to 266 points and the higher the score the better the functionality.

SECONDARY OUTCOMES:
Muscle strength | Baseline, after 3 weeks and after 6 weeks.
  The change in muscle strength will be assessed by the Medical Research Council (MRC) scale and by test of maximum repetition (1RM)
Quadriceps muscle thickness | Baseline and after 6 weeks
  The change in quadriceps muscle thickness will be evaluated for the acquisition of ultrasound images using a high resolution ultrasound device (Vivid-i, GE, USA). In order to verify the thickness of the muscle, the distance between the superficial and deep aponeurosis is measured.The thickness is given in centimeters.
Echogenicity of the rectus femoris muscle | Baseline and after 6 weeks
  The change in echogenicity will be evaluated for the acquisition of ultrasound images of the rectus femoris muscle using a high resolution ultrasound device (Vivid-i, GE, USA). To check the echogenicity of the rectus femoris an image of the cross-sectional area of the muscle will be taken. The echogenicity measurement is given in an arbitrary unit.
Spasticity | Baseline, after after 3 weeks and after 6 weeks
  The change in spasticity will be assessed by the Modified Ashworth Scale. This scale consists of an ordinal classification of 5 points for grading the resistance found during passive stretching, with 0 indicating normal muscle tone and 4 severe increase in tone. The higher the score, the greater the spasticity.
Mobility | After 3 weeks and after 6 weeks
  The change in mobility will be assessed using the Timed Up and Go test (TUG), which will be associated with an inertial sensor
Disability and dependence | Baseline and after 6 weeks
  The change in disability and dependency will be assessed using the Modified Rankin Scale. This instrument has 6 scores, where: 0 = asymptomatic; 1 = symptoms without disabilities; 2 = mild disability; 3 = moderate disability; 4 = moderate to severe disability; 5 = severe disability and 6 = death. The higher the score, the greater the degree of disability and dependence.
Quality of life indicator | Baseline and after 6 weeks
  The change in quality of life will be assessed using the EuroQol-5D questionnaire. This is a generic instrument that assesses mobility, personal care, usual activities, pain and anxiety/depression. It allows to generate a global index of the value of an individual's health status. The number 1 indicates the best state of health (perfect health) and 0 the worst state of health (death).
Heart rate | From the 1st to the 18th day/session
  Heart rate will be assessed by pulse oximetry
Peripheral arterial oxygen saturation | From the 1st to the 18th day/session
  Peripheral arterial oxygen saturation will be assessed by pulse oximetry
Systolic blood pressure | From the 1st to the 18th day/session
  Systolic blood pressure will be assessed through sphygmomanometer
Diastolic blood pressure | From the 1st to the 18th day/session
  Diastolic blood pressure will be assessed through sphygmomanometer
Muscle pain | From the 1st to the 18th day/session
  Pain perception will be assessed using the Visual Analog Scale. This scale ranges from 0 to 10, where 0 indicates no pain and 10 maximum pain.
Lower limb fatigue | From the 1st to the 18th day/session
  Lower limb fatigue will be assessed by Borg effort subjective perception scale. This scale ranges from 0 to 10, where 0 indicates no effort or fatigue and 10 indicates maximum effort.
Time of hospital stay | From the 1st to the last day of hospitalization
  The days between admission and hospital discharge will be counted

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo DM Plentz, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre